CLINICAL TRIAL: NCT02521181
Title: The BASE Study: Bicarbonate Administration to Stabilize eGFR
Brief Title: The BASE Study: Bicarbonate Administration to Stabilize Estimated Glomerular Filtration Rate (eGFR)
Acronym: BASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jennifer Gassman, PhD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Jennifer Gassman, PhD, Principal Investigator-Data Coordinating Center, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DK099877-B; U01DK099877 (NIH)
Record Dates: First submitted 2015-04-27; First posted 2015-08-13 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lower Dose Sodium Bicarbonate (Experimental): Participants will receive oral 0.5 milliequivalents (mEq)/kg-lean body weight (LBW)/day of sodium bicarbonate. Half of the total daily dose is taken in the morning and the other half is taken in the evening. (If the number of capsules is an odd number, the greater number of capsules will be taken in the morning.)
  Interventions: Drug: Lower Dose Sodium Bicarbonate
- Higher Dose Sodium Bicarbonate (Experimental): Participants will receive 0.8 mEq/kg-LBW/day of sodium bicarbonate. Half the total daily dose is taken in the morning and the other half is taken in the evening. (If the number of capsules is an odd number, the greater number of capsules will be taken in the morning.)
  Interventions: Drug: Higher Dose Sodium Bicarbonate
- Placebo (Placebo Comparator): Participants will take the same number of placebo capsules as if they were assigned to receive either 0.5 mEq/kg-LBW/day or 0.8 mEq/kg-LBW/day of sodium bicarbonate. Half the total daily dose is taken in the morning and the other half is taken in the evening. (If the number of capsules is an odd number, the greater number of capsules will be taken in the morning.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lower Dose Sodium Bicarbonate — Lower dose oral Sodium Bicarbonate (0.5 milliequivalents (mEq)/kg-LBW/day)
  Arms: Lower Dose Sodium Bicarbonate
Drug: Higher Dose Sodium Bicarbonate — Higher dose oral Sodium Bicarbonate (0.8 mEq/kg-LBW/day)
  Arms: Higher Dose Sodium Bicarbonate
Drug: Placebo — Oral placebo equivalent to either 0.5 mEq/kg-LBW/day or 0.8 mEq/kg-LBW/day of Sodium Bicarbonate
  Arms: Placebo

SUMMARY:
The two doses of sodium bicarbonate being tested are 0.5 and 0.8 mEq/kg-lean body weight (LBW) per day. Sodium bicarbonate, also known as baking soda, may help prevent kidney failure in people with chronic kidney disease. However, the dose to prescribe in order to test this possibility in a clinical trial is uncertain. The BASE pilot clinical trial will help determine the best dose of sodium bicarbonate to prescribe in a future study that will test the long-term safety and efficacy of sodium bicarbonate as a treatment to preserve kidney function in individuals with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Serum bicarbonate 20-28 mEq/L at screening (the average of the two most recent values in Baseline must be 20-28 mEq/L prior to randomization)
2. Moderate to severe chronic kidney disease (CKD) at the time of screening, defined as one of the following:

   * eGFR 20-44 ml/min/1.73m2 or
   * eGFR 45-59 ml/min/1.73m2 plus random urinary albumin:creatinine (ACR) ≥100 mg/gm
3. Blood pressure <160/100 mm Hg at screening (must be <150/100 mm Hg prior to randomization)
4. Lean body weight 38.0-96.0 kg at the time of screening
5. Age allowing legal consent without parental involvement (18-21 years, depending on individual state regulations)
6. Able to provide consent
7. Able to travel to study visits
8. Able to read English
9. In the opinion of the site investigator, willing and able to follow the study treatment regimen and comply with the site investigator's recommendations
10. In the opinion of the site investigator, medically stable

Exclusion Criteria:

1. Use of chronic daily oral alkali (such as sodium bicarbonate, sodium citrate, potassium citrate, etc) with one exception: calcium carbonate ≤1500 mg/day is allowed, as some will take this for the indication of bone health
2. On five or more antihypertensive and/or diuretic agents, regardless of the indication
3. Serum potassium <3.3 or ≥5.5 mEq/L at screening (must be 3.5-5.5 mEq/L prior to randomization)
4. Self-reported vegetarian
5. New York Heart Association Class 3 or 4 heart failure symptoms, known left ventricular ejection fraction ≤30%, or hospital admission for heart failure within the past 3 months
6. Frequent urinary tract infections (≥2 in the past year)
7. Presence of indwelling urinary catheter or urinary conduit (such as neobladder or urostomy)
8. Factors judged to limit adherence to interventions (e.g., alcoholism, history of missing clinic visits, chronic gastrointestinal disorder that makes compliance with the intervention unreliable)
9. Organ transplant recipients (excluding cornea)
10. Active glomerular disease requiring or potentially requiring immunosuppressive treatment
11. Chronic immunosuppressive therapy (for ≥3 months) for any indication. This does not include oral steroids <10 mg per day, inhaled steroids, or topical steroids
12. Anticipated initiation of dialysis or kidney transplantation within 12 months as assessed by the site investigator
13. Current participation in another interventional research study
14. Malignancy requiring therapy within 2 years (basal or squamous cell skin carcinoma and localized prostate cancer are exempted)
15. Pregnancy or planning to become pregnant or currently breast-feeding. Women of childbearing potential (pre-menopausal and not surgically sterilized) will have urine pregnancy test before enrollment.
16. Life expectancy <12 months as determined by the site investigator
17. Institutionalized individuals, including prisoners and nursing home residents
18. Plans to leave the immediate area within the next 12 months
19. Routinely leaves town for multiple weeks each year such that protocol visits would be missed
20. Chronic use of supplemental oxygen
21. Use of both angiotensin-converting-enzyme inhibitor (ACEI) and Angiotensin II Receptor Blockers (ARBs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Flessner, MD, PhD, Study Director — DKUHD, NIDDK, NIH; John W. Kusek, PhD, Study Director — DKUHD, NIDDK, NIH; Linda Fried, MD, MPH, Study Chair — VA Pittsburgh Healthcare System
Locations (7):
- United States (7):
  - Denver Nephrology Research, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Data Coordinating Center; Cleveland Clinic Foundation; Quantitative Health Sciences; 9500 Euclid Avenue, Cleveland, Ohio
  - Baylor/Scott & White, Temple, Texas
  - University of Utah, Salt Lake City, Utah
  - Utah VA, Salt Lake City, Utah

REFERENCES:
- [Derived] Raphael KL, Katz R, Larive B, Kendrick C, Isakova T, Sprague S, Wolf M, Raj DS, Fried LF, Gassman J, Hoofnagle A, Cheung AK, Ix JH. Oral Sodium Bicarbonate and Bone Turnover in CKD: A Secondary Analysis of the BASE Pilot Trial. J Am Soc Nephrol. 2024 Jan 1;35(1):57-65. doi: 10.1681/ASN.0000000000000264. Epub 2023 Dec 4. PMID 38170601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the CKD medical clinic patients of the recruiting centers.
Period: Overall Study
Arm/Group | Lower Dose Sodium Bicarbonate | Higher Dose Sodium Bicarbonate | Placebo
Started | 52 | 90 | 52
Completed | 52 (All patients included in primary analysis) | 90 (All patients included in primary analysis) | 52 (All patients included in primary analysis)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Dose Sodium Bicarbonate | Higher Dose Sodium Bicarbonate | Placebo | Total
Number analyzed (Participants) | 52 | 90 | 52 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 39 | 15 | 74
  >=65 years | 32 | 51 | 37 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (14.0) | 67.3 (10.8) | 66.2 (10.8) | 66.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 13 | 63
  Male | 31 | 61 | 39 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 3 | 17
  Not Hispanic or Latino | 46 | 82 | 49 | 177
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 17 | 27 | 23 | 67
  White | 28 | 55 | 26 | 109
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 52 | 90 | 52 | 194
CKD Stage [Count of Participants; unit: Participants]
  Stage 3A (eGFR 45-60) | 9 | 17 | 4 | 30
  Stage 3B (eGFR 30-45) | 30 | 46 | 31 | 107
  Stage 4 (eGFR 15-30) | 13 | 27 | 17 | 57
Diabetes Mellitus [Count of Participants; unit: Participants] | 27 | 53 | 25 | 105
History of Heart Disease [Count of Participants; unit: Participants] | 18 | 28 | 20 | 66
Congestive Heart Failure [Count of Participants; unit: Participants] | 5 | 8 | 7 | 20
COPD [Count of Participants; unit: Participants] | 4 | 6 | 0 | 10
Smoking Status [Count of Participants; unit: Participants]
  Never | 26 | 47 | 25 | 98
  Former Smoker | 15 | 39 | 25 | 79
  Current Smoker | 11 | 4 | 2 | 17
Weight [Mean (Standard Deviation); unit: kg] | 96.1 (25.8) | 95.4 (22.4) | 93.6 (20.3) | 95.1 (22.7)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.8 (8.43) | 32.8 (7.87) | 31.6 (5.92) | 32.5 (7.54)
Lean Body Mass [Mean (Standard Deviation); unit: kg] | 58.4 (10.7) | 58.4 (9.84) | 58.7 (9.44) | 58.5 (9.91)
Systolic BP [Mean (Standard Deviation); unit: mm Hg] | 127 (13.7) | 127 (12.3) | 127 (13.0) | 127 (12.8)
Ace/ARB Use [Count of Participants; unit: Participants] | 40 | 60 | 35 | 135
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 36.5 (9.56) | 36.4 (9.60) | 34.5 (8.59) | 35.9 (9.32)
Urine Albumin / Creatinine Ratio [Median (Inter-Quartile Range); unit: g/mg] | 222 [57.8 to 788] | 176 [22.9 to 769] | 147 [12.2 to 593] | 181 [24.9 to 745]
Serum Bicarbonate [Mean (Standard Deviation); unit: meq/L] | 24.2 (2.25) | 24.2 (2.38) | 23.8 (2.17) | 24.1 (2.28)
Serum Potassium [Mean (Standard Deviation); unit: meq/L] | 4.5 (0.4) | 4.4 (0.4) | 4.5 (0.5) | 4.5 (0.4)
Urinary Ammonium [Mean (Standard Deviation); unit: mmol/day] | 19.3 (10.5) | 22.0 (12.2) | 20.5 (13.2) | 20.9 (12.0)
Urinary PH [Mean (Standard Deviation); unit: units on a scale] | 5.86 (0.46) | 5.75 (0.46) | 5.81 (0.56) | 5.80 (0.49)
Estimated DIetary Protein Intake [Mean (Standard Deviation); unit: g/day] | 73.3 (25.4) | 81.9 (30.5) | 79.1 (29.5) | 78.8 (29.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Dose Arm Prescribed (i) Full Randomized Sodium Bicarbonate Dose at End of 28 Weeks & (ii) at Least 25% of Randomized Sodium Bicarbonate Dose at End of 28 Weeks as a Proportion of the Number Randomized to That Group
Description: The prescribed dose for each participant at the end of 28 weeks will be determined by the safety and tolerability of each dose during the intervention period. The primary assessments will examine the percentage of participants in each dose arm who are prescribed (i) the full randomized sodium bicarbonate dose according to the protocol at the end of 28 weeks and (ii) at least 25% of the randomized sodium bicarbonate dose according to the protocol at the end of 28 weeks. The two doses of sodium bicarbonate being tested are 0.5 and 0.8 mEq/kg-lean body weight per day.
Time Frame: Baseline, 28 weeks
Measure: Number; unit: participants
Arm/Group | Lower Dose Sodium Bicarbonate | Higher Dose Sodium Bicarbonate | Placebo
Number analyzed (Participants) | 52 | 90 | 52
participants
  Number of Patients Completing on Full Dose | 50 | 78 | 45
  Num of Patients Completing on >= 25% of Full Dose | 51 | 82 | 48

ADVERSE EVENTS:
Time Frame: 32 Weeks
Arm/Group | Lower Dose Sodium Bicarbonate | Higher Dose Sodium Bicarbonate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/90 | 1/52
Serious Adverse Events (participants affected / at risk) | 5/52 | 16/90 | 7/52
Other Adverse Events (participants affected / at risk) | 40/52 | 74/90 | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Sodium Bicarbonate (N=52) | Higher Dose Sodium Bicarbonate (N=90) | Placebo (N=52)
Reached ESRD (Dialysis or Transplant) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular Hospitalizations (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Gastrointestinal Hospitalizations (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Infection Hospitalizations (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2)
Renal Hospitalizations (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Malignancy Hospitalizations (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Injury Hospitalizations (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Respiratory Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal Hospitalizations (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 0 (0)
Endocrine Disorder Hospitalizations (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular Hospitalizations (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Psychiatric Hospitalizations (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Sodium Bicarbonate (N=52) | Higher Dose Sodium Bicarbonate (N=90) | Placebo (N=52)
Severe gastrointestinal symptoms (Gastrointestinal disorders) | 9 (15) | 16 (28) | 5 (6) — Highest level of symptoms was severe
Moderate gastrointestinal symptoms (Gastrointestinal disorders) | 7 (17) | 22 (36) | 13 (17) — Highest level of symptoms is moderate
Mild gastrointestinal symptoms (Gastrointestinal disorders) | 24 (54) | 36 (107) | 24 (62) — Highest level of symptoms is mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT02521181/Prot_SAP_000.pdf